CLINICAL TRIAL: NCT05993364
Title: Role of Expiratory Flow Acceleration in the Management of Bronchial Secrections in Severe Acquired Brain Injury: a Pilot Randomized Controlled Study
Brief Title: Efficacy of EFA in Acquired Brain Injury
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Fondazione Don Carlo Gnocchi Onlus (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: EFA-ABI
Record Dates: First submitted 2023-08-07; First posted 2023-08-15 (Actual); Last update posted 2024-08-09 (Actual); Status verified 2024-08

CONDITIONS: Acquired Brain Injury; Comparative Effectiveness Research; Lung Diseases, Obstructive
Keywords: Expiratory Flow Accelerator; Tracheobronchial secretions; Tracheobronchial clearance; Airways clearance; Pulmonary infections; Pulmonary obstruction; Decannulation; Tracheal cannula; Effectiveness; Acquired Brain Injury; Controlled study
MeSH Terms: conditions — Brain Injuries; Lung Diseases, Obstructive; Airway Obstruction

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control group (Active Comparator): The control group receive a standard rehabilitative treatment to improve the secretions management and the respiratory function. Besides, the control group receives a traditional rehabilitative treatment carried out by the speech and language pathologist.
  Interventions: Device: In-Exufflator Machine; Other: Traditional respiratory treatment; Other: Traditional swallowing treatment
- Experimental group (Experimental): The experimental group receives the same standard rehabilitative treatment performed with the control group. In addition, sessions with the EFA technology are provided.
  Interventions: Device: Free Aspire with Expiratory Flow Accelerator (EFA) technology; Device: In-Exufflator Machine; Other: Traditional respiratory treatment; Other: Traditional swallowing treatment

INTERVENTIONS:
Device: Free Aspire with Expiratory Flow Accelerator (EFA) technology — Treatment sessions during which the EFA technology is used. Depending on the patient's clinical conditions, an oxygen additional support can be provided, while using the device. If present, during the sessions the tracheal cannula must be cuffed. Tracheal cannula aspiration must be provided when necessary. Sessions take place three times a day and take 20 minutes each time, from Monday to Saturday.
  Arms: Experimental group
Device: In-Exufflator Machine — Sessions using the In-Exufflator machine to improve the cough function, when the oxygen saturation decreases and the bronchial secretions increases.
Other: Traditional respiratory treatment — Standard rehabilitative treatment to improve the secretions management, that includes:
  * A change of the patient posture every three hours;
  * Airways humidification depending on the secretions features;
  * Aspiration in the tracheal cannula whenever necessary.
Other: Traditional swallowing treatment — Traditional rehabilitative treatment carried out by the speech and language pathologist in order to:
  * Obtain decannulation (when a tracheal cannula is applied) following the Bargellesi Protocol steps;
  * Improve oral structures strength and motility;
  * Improve oral and perioral sensitivity with thermal or gustative or tactile stimulations;
  * Improve the swallowing function with food trials of different consistencies, volume and temperature;
  * Improve swallow efficacy and safety through the prescription of compensatory postures;

SUMMARY:
Acquired brain injury (ABI) is one of the biggest cause of death and disability in the world. Patients with ABI often have difficulties with swallow and breath.

The study purpose is to evaluate if the Expiratory Flow Accelerator (EFA) technology has positive effects on the respiratory and swallowing function in patients with acquired brain injury (ABI). Researchers recruit patients at Centro Ettore Spalenza-Fondazione Don Carlo Gnocchi in Rovato, Italy.

To partecipate, patients should satisfy certain eligibility criteria; they will not be enrolled if they satisfy exclusion criteria.

If a patient can be recruited, researchers conduct the baseline assessment lasting 1 one week. After that, the patient will be randomized to the study or control group. If the patient is in the control group, he will receive a traditional rehabilitation treatment. Otherwise, the patient will receive an additional treatment with the EFA device.

Researchers will assess again the patient (with the same procedures of baseline assessment) after 8 weeks of treatment. They want to see if the EFA device could help patients with ABI to improve their health conditions.

DETAILED DESCRIPTION:
Acquired Brain Injury (ABI) is one of the most frequent cause of death and disability worldwide. Swallowing disorders and cough insufficiency followed by pulmonary infections and a bad secretions management are some of the associated complications. When a tracheal cannula is applied, the patient conditions could get worse. Unfortunately ABI patients often can't properly collaborate to the treatment/assessment processes due to their consciousness disorders. According to all these reasons, ABI patients need a multi-professional assistance focused on swallowing and respiratory rehabilitative treatments to improve their health conditions.

Free Aspire device with Expiratory Flow Accelerator (EFA) technology, thanks to the expiratory flow acceleration, allows to remove tracheobronchial secretions and an improvement of the swallowing ability.

EFA, compared to other devices, is simple to use and does not require the active collaboration of the patient. Indeed, the purpose of the study is to investigate its effects on secretion management ability and to evaluate if EFA can reduce the frequency of Hospital Acquired Pneumonia (HAP). In addition, the study evaluates the effectiveness of EFA in accelerating tracheotomy weaning.

Patients will be recruited following accurate inclusion/exclusion criteria at Centro Ettore Spalenza-Fondazione Don Carlo Gnocchi in Rovato, Italy.

At baseline assessment (1 week), the following parameters will be assessed daily for each patient recruited:

* Saturation of Peripheral Oxygen (Sp02)
* Oxygen supply as fraction of inspired oxygen (Fi02)
* Number of oxyhemoglobin desaturation episodes.
* Number of the needed aspiration in the tracheal cannula due to tracheo-bronchial obstruction.
* Number of and duration of antibiotic therapy courses due to HAP.

After baseline evaluation, patients will be randomized to the control or to the experimental group.

Every patient undergoes the same evaluation during the 8 weeks of treatment. Additionally, an arterial blood gas analysis will be performed every week for clinically monitoring the patients recruited.

The control group receives standard rehabilitation treatments carried out by physical therapists and speech and language pathologists. This treatment takes place every day (from Monday to Saturday) in daily sessions that lasts from 30 to 60 minutes each.

In addition to that, the experimental group undergoes treatment sessions using Free Aspire Device with Expiratory Flow Accelerator (EFA) technology, three times a day from Monday to Friday and one time a day on Saturday. The sessions last 20 minutes each. EFA technology generates a non invasive expiratory flow acceleration, allowing the bronchial secretions removal without requiring the active collaboration of the patient. EFA could be applied through the tracheal cannula, a facial mask or a mouthpiece.

Both the control and the experimental treatments last 8 weeks. Researchers expect that the experimental group shows an improvement of the tracheo-bronchial clearance and of the respiratory and swallowing functions. As a result, there should be fewer episodes of desaturation and HAP and less need for tracheal aspirations. In addition, patients with tracheal cannula should show earlier decannulation..

Researchers want to prove that EFA could be an effective and simple device to use in the rehabilitation of patients with ABI, available to the entire multi-professional equipe, caregivers included.

ELIGIBILITY:
Inclusion Criteria:

* Age higher than 18 years old;
* Hospitalization after diagnosis of Acquired Brain Injury (both traumatic and vascular)
* Levels of Cognitive Functioning Scale (LCFS) score between 1and 5;
* Presence of spontaneous breathing, at least during the day

Exclusion Criteria:

* Need of mechanical ventilation for more than 12 hours a day;
* Presence of tracheal stoma not properly healed after the removal of the tracheal cannula.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2024-02-19 (Actual); Primary Completion 2025-02 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Change of oxyhemoglobin desaturation episodes | During the data collection in the 8 weeks of treatment for each patient, the number of oxyhemoglobin desaturation episodes will be registered
  Change in the the frequency of oxyhemoglobin desaturation episodes.

SECONDARY OUTCOMES:
Reduction of tracheal cannula aspiration | During the data collection in the 8 weeks of treatment for each patient, the number of tracheal cannula aspiration will be registered.
  Reduction of the number of the needed aspiration in the tracheal cannula due to tracheo-bronchial obstruction
Number of patient that develop hospital-acquired pneumonia | During the data collection in the 8 weeks of treatment for each patient, the number of hospital-acquired pneumonia that require an antibiotic treatment will be registered
  Variation in the number of cases of hospital-acquired pneumonia.
Change of tracheostomy weaning time | From baseline to last observation (at the of 8 weeks treatment)
  Change of time need to accomplish tracheostomy weaning, measured in days
Staff satisfaction | From baseline to last observation (at the of 8 weeks treatment)
  A 5 point Likert scale will be administered to rehabilitation staff about the ease of use of the EFA device and the time expenditure. Score from 0 (minimum value) to 4 (maximum value).

CONTACTS AND LOCATIONS:
Overall Officials: Luca NC Bianchi, MD, Principal Investigator — IRCSS Fondazione Don Carlo Gnocchi
Locations (1):
- Fondazione Don Carlo Gnocchi - Centro Ettore Spalenza, Rovato, BS, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ahmed S, Venigalla H, Mekala HM, Dar S, Hassan M, Ayub S. Traumatic Brain Injury and Neuropsychiatric Complications. Indian J Psychol Med. 2017 Mar-Apr;39(2):114-121. doi: 10.4103/0253-7176.203129. PMID 28515545
- [Background] Belli S, Cattaneo D, D'Abrosca F, Prince I, Savio G, Balbi B. A pilot study on the non-invasive management of tracheobronchial secretions in tracheostomised patients. Clin Respir J. 2019 Oct;13(10):637-642. doi: 10.1111/crj.13074. Epub 2019 Aug 26. PMID 31390146
- [Background] Borders JC, Gibson AL, Grayev A, Thibeault S. Predictors of dysphagia in critically injured patients with neck trauma. J Crit Care. 2018 Apr;44:312-317. doi: 10.1016/j.jcrc.2017.12.004. Epub 2017 Dec 7. PMID 29268199
- [Background] Bone DK, Davis JL, Zuidema GD, Cameron JL. Aspiration pneumonia. Prevention of aspiration in patients with tracheostomies. Ann Thorac Surg. 1974 Jul;18(1):30-7. doi: 10.1016/s0003-4975(10)65714-1. No abstract available. PMID 4834725
- [Background] Cook AM, Peppard A, Magnuson B. Nutrition considerations in traumatic brain injury. Nutr Clin Pract. 2008 Dec-2009 Jan;23(6):608-20. doi: 10.1177/0884533608326060. PMID 19033220
- [Background] Eskildsen SJ, Jakobsen D, Riberholt CG, Poulsen I, Curtis DJ. Protocol for a scoping review study to identify and map treatments for dysphagia following moderate to severe acquired brain injury. BMJ Open. 2019 Jul 17;9(7):e029061. doi: 10.1136/bmjopen-2019-029061. PMID 31320355
- [Background] Farneti D. Pooling score: an endoscopic model for evaluating severity of dysphagia. Acta Otorhinolaryngol Ital. 2008 Jun;28(3):135-40. PMID 18646575
- [Background] Galeoto G, Turriziani S, Berardi A, Sansoni J, Santilli V, Mascio M, Paoloni M. Levels of Cognitive Functioning Assessment Scale: Italian cross-cultural adaptation and validation. Ann Ig. 2020 Jan-Feb;32(1):16-26. doi: 10.7416/ai.2020.2326. PMID 31713573
- [Background] Lanini B, Binazzi B, Romagnoli I, Chellini E, Pianigiani L, Tofani A, Molino Lova R, Corbetta L, Gigliotti F. Tracheostomy decannulation in severe acquired brain injury patients: The role of flexible bronchoscopy. Pulmonology. 2023 Dec;29 Suppl 4:S80-S85. doi: 10.1016/j.pulmoe.2021.05.006. Epub 2021 Jul 2. PMID 34219041
- [Background] Ninfa A, Pizzorni N, Eplite A, Moltisanti C, Schindler A. Validation of the Italian Version of the Functional Oral Intake Scale (FOIS-It) Against Fiberoptic Endoscopic Evaluation of Swallowing and Nutritional Status. Dysphagia. 2022 Feb;37(1):137-147. doi: 10.1007/s00455-021-10257-9. Epub 2021 Feb 16. PMID 33591464
- [Background] Patrizio G, D'Andria M, D'Abrosca F, Cabiaglia A, Tanzi F, Garuti G, Nicolini A. Airway Clearance with Expiratory Flow Accelerator Technology: Effectiveness of the "Free Aspire" Device in Patients with Severe COPD. Turk Thorac J. 2019 Jul 30;20(4):209-215. doi: 10.5152/TurkThoracJ.2018.18053. Print 2019 Oct. PMID 31390330
- [Background] Riboldazzi G, Spinazza G, Beccarelli L, Prato P, Grecchi B, D'Abrosca F, Nicolini A. Effectiveness of expiratory flow acceleration in patients with Parkinson's disease and swallowing deficiency: A preliminary study. Clin Neurol Neurosurg. 2020 Dec;199:106249. doi: 10.1016/j.clineuro.2020.106249. Epub 2020 Sep 28. PMID 33039853
- [Background] Rosenbek JC, Robbins JA, Roecker EB, Coyle JL, Wood JL. A penetration-aspiration scale. Dysphagia. 1996 Spring;11(2):93-8. doi: 10.1007/BF00417897. PMID 8721066
- [Background] Rotolo N, Cattoni M, D'Andria M, Cavanna L, Patrizio G, Imperatori A, Nicolini A. Comparison of an expiratory flow accelerator device versus positive expiratory pressure for tracheobronchial airway clearance after lung cancer lobectomy: a preliminary study. Physiotherapy. 2021 Mar;110:34-41. doi: 10.1016/j.physio.2019.01.011. Epub 2019 Jan 26. PMID 33563372
- [Background] Thomas-Stonell N, Greenberg J. Three treatment approaches and clinical factors in the reduction of drooling. Dysphagia. 1988;3(2):73-8. doi: 10.1007/BF02412423. No abstract available. PMID 3271655
- [Background] Ward EC, Green K, Morton AL. Patterns and predictors of swallowing resolution following adult traumatic brain injury. J Head Trauma Rehabil. 2007 May-Jun;22(3):184-91. doi: 10.1097/01.HTR.0000271119.96780.f5. PMID 17510594
- See also: Bargellesi Protocol — https://www.minervamedica.it/en/journals/medicina-riabilitativa/article.php?cod=R47Y2013N01A0009
- See also: Cranial Nerve Examination for Neurogenic Dysphagia Patients-I&I Test — https://www.omicsonline.org/open-access-pdfs/cranial-nerve-examination-for-neurogenic-dysphagia-patients-2161-119X-1000319.pdf